CLINICAL TRIAL: NCT06436794
Title: "Mantou" Screening for Gestational Diabetes Mellitus Before 20 Weeks of Gestation:A Prospective,Multicenter Study.
Brief Title: "Mantou" Screening for GDM Before 20 Weeks of Gestation
Status: Not yet recruiting | Type: Observational
Sponsor: Jiang Ziyan (Other)
Responsible Party: Sponsor-Investigator, Jiang Ziyan, MD, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Other Study IDs: MS-GDM-01
Record Dates: First submitted 2024-04-16; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: GDM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 12-14 weeks
- 15-17 weeks
- 18-20 weeks

SUMMARY:
Gestational diabetes mellitus (GDM) can occur in overweight, hyperinsulinemia, insulin resistance pregnant women, or lean, insulin deficiency pregnant women. At least 5% of all pregnant women will develop GDM, which is even higher among Asians. Poor control of GDM in late pregnancy will increase the following risks: macrosomia, preeclampsia, shoulder dystocia, cesarean section, stillbirth and other risks. At present, the screening method for GDM is 75g of glucose OGTT test. However, when drinking sugared water on an empty stomach, the pregnant women will feel nausea, stomach burning, and hunger when waiting for blood drawing. Some women vomit after drinking sugared water, resulting in inaccurate test results and poor compliance, affecting the accuracy of diagnosis of GDM. "Sugar tolerance Mantou" has been used for screening diabetes since 1982. It is made of 100g flour and contains 75g glucose of the same amount. It is a feasible method to use Mantou instead of sugar powder to screen GDM. Mantou is an acceptable diet for Chinese people, which greatly reduces nausea, vomiting, hunger and other discomfort, and increases GDM screening rate. At present, the cesarean section rate in China remains high, and the weight and nutritional management of pregnant women are not satisfied. Many pregnant women, especially those in country-level areas, have already gained excessive weight when referred from to delivery hospitals, leading to an increase in pregnancy complications such as preeclampsia and macrosomia, increasing the cesarean section rate and delivery risk. Therefore, it is necessary to screen GDM in advance. Moving forward the screening of GDM and strengthening the management of pregnant women's weight can effectively reduce the occurrence of pregnancy complications.

ELIGIBILITY:
Inclusion Criteria:Singleton , before 20 weeks of gestation, aged 18-40 years old, able to understand the experimental requirements, willing and able to follow the experimental and follow-up procedures.

Exclusion Criteria: diabetes diagnosed before pregnancy, serious heart disease, blood disease, immune system disease and other unsuitable for pregnancy, twin or multiple pregnancy, age<18 or>40, fetal death in utero before 28 weeks, serious mental illness, and inability to communicate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant woman
Sampling Method: Non-Probability Sample
Enrollment: 5925 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
GDM incidence rate | up to 28 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided